CLINICAL TRIAL: NCT02433964
Title: EVALUATION OF THERAPEUTIC EFFECTS OF LED (627 +/- 10nm) THE INITIAL PHASE OF THE ANKLE SPRAINS TREATMENT - A RANDOMIZED PLACEBO-CONTROLLED CLINICAL TRIAL
Brief Title: Evaluation of Therapeutic Effects of LED (627 +/- 10nm) The Initial Phase of the Ankle Sprains Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: University of Vale of Paraíba
Record Dates: First submitted 2015-04-01; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Ankle Sprain
Keywords: laser; LED; PRICE; pain; edema
MeSH Terms: conditions — Ankle Injuries; Pain; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LED group (Experimental): Treated by a device LED - LED: power 60mW, 627nm wavelength ± 10nm and 1,3cm2 beam output. The energy density used was 10J / cm2 with time of 2 minutes and 47 seconds per flash of the beam, which is unique for each ten points in the lateral region of the ankle edema. The volunteers underwent previous cleaning application points with cotton soaked in 70% alcohol, positioned for high stretcher in the supine position and wearing goggles. The LED was applied in a timely manner, wherein the skin contact surfasse at an angle of 90 °, the ten points were irradiated in a 1cm2 area selected by a single investigator. One session was performed every 24 hours for six consecutive days. Ice applications were made associated with semi-rigid compression bandage, with the patient lying supine and the affected limb in elevation under a foam wedge in the same period.
  Interventions: Other: Grupo LED
- Placebo group (Placebo Comparator): Both volunteers LED group and the placebo group were treated with the same procedure, with the LED device in the placebo group remained off.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Grupo LED
  Arms: LED group
Other: Placebo — ledterapia off + price
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the therapeutic effects of the LED (627 +/- 10 nm) with respect to the localized pain and local swelling of ankle sprains in the initial phase.

DETAILED DESCRIPTION:
A variety of therapies for the treatment of sprains has emerged as they occur advances in technological applications. Therapy with coherent and non-coherent light is a treatment modality for a variety of musculoskeletal injuries. The main benefits certificates for phototherapy are the reduction of nociceptive processes, tissue remodeling, among others. The aim of the present paper is to analyze the changes caused by the use of LED (627 +/- 10 nm) with an energy density of 10 J / cm2 in 40 subjects divided into two groups (placebo and LED). All volunteers participating in this study had ankle inversion sprain grade II treated with the price technique. The study was performed in six days. And the results were verified by review of all individuals, through the Visual Analogue Scale (VAS) of pain, McGill Pain Questionnaire and Titrimetry. Measurements were performed at first, third and sixth day's of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Active individuals
* With medical referral
* With clinical diagnosis of inversion sprain grade II
* The day he suffered the injury
* Without prescriptions

Exclusion Criteria:

* Individuals who had previous trauma and orthopedic disorders such as fractures, tendinopathy, previous surgical procedure
* Other systemic diseases.

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
edema, measured by volumetry | the development of edema in 6 days
  Edema was measured on the first, third and sixth day

SECONDARY OUTCOMES:
pain, measured by the Visual Analogue Pain Scale (VAS) and McGill Pain Questionnaire | the evolution of the pain in 6 days
  Pain was measured on the first, third and sixth day

CONTACTS AND LOCATIONS:
Overall Officials: Bruno de Moraes Prianti, Principal Investigator — Universidade do Vale do Paraíba
Locations (1):
- Lasertherapy and Photobiology Center, São José dos Campos, São Paulo, Brazil